CLINICAL TRIAL: NCT06040450
Title: The Impact of Outdoor Sports Practice on the Well-Being of Disabled People : a Cross-Sectional Study
Brief Title: The Impact of Outdoor Sports Practice on the Well-Being of Disabled People
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut de Sante Parasport Connecte Synergies (Other)
Collaborators: Fédération Française Handisport (FFH) (Unknown); Université de Montpellier - UMR Santé, Education et Situations de Handicap (SANTESIH) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2023-004
Record Dates: First submitted 2023-09-07; First posted 2023-09-15 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Disability or Chronic Disease Leading to Disablement
Keywords: Physical activities, Outdoor sports, Disability
MeSH Terms: conditions — Motor Activity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- All subjects with impairments
  Interventions: Other: Questionnaire survey
- All subjects without impairments
  Interventions: Other: Questionnaire survey

INTERVENTIONS:
Other: Questionnaire survey — On outdoor sports practice activity, barriers to practice, impacts on well-being.

SUMMARY:
Survey of the members of the French Handisports Federation (FFH) practicing outdoor sports.

DETAILED DESCRIPTION:
This is a national cross-sectional study to investigate the impact of outdoor sports practice on the well-being and self-esteem of people with disabilities.

The study is based on a survey of FFH members practicing outdoor sports. The survey will be distributed between October and November 2023 via the federation's internal communication system. Data will be collected on outdoor sports activity, psychological impact and barriers to practice.

Analyses will be made between able-bodied and disabled members, between types of disability, and between types of outdoor sport practiced (water, land and air).

Analysis will be based on anomysed data and will respect the MR004 methodology.

ELIGIBILITY:
Inclusion Criteria:

* Being a member of the French Handisport Federation between September 2022 and August 2023
* Practicing outdoor sports

Exclusion Criteria:

* Persons who have objected to be contacted by e-mail

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Members of the French Handisport Federation practicing outdoor sports
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Impact of my outdoor sports on my well-being | Baseline
  Rating Scale : 1 (low) to 10 (high)

SECONDARY OUTCOMES:
Impact of my outdoor sports on my self-esteem | Baseline
  Rating Scale : 1 (low) to 10 (high)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent T. Carpentier, MD-MSc, Study Director — Institut de Sante Parasport Connecte Synergies; Eric Perera, PhD, Study Director — Montpellier University - SANTESIH; Emmanuel Buchoud, Study Director — French Handisport Federation
Locations (1):
- French Handisport Federation, Paris, France

IPD SHARING:
Plan to Share IPD: No